CLINICAL TRIAL: NCT05017935
Title: RADIANCE Continued Access Protocol (RADIANCE CAP): A Study of the ReCor Medical Paradise System in Clinical Hypertension
Brief Title: RADIANCE Continued Access Protocol
Acronym: RADIANCE CAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ReCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-0932
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Hypertension; Hypertension, Resistant to Conventional Therapy; Vascular Diseases; Cardiovascular Diseases
Keywords: Blood Pressure; Uncontrolled Hypertension; Essential Hypertension; Resistant Hypertension; Denervation
MeSH Terms: conditions — Hypertension; Hypertension Resistant to Conventional Therapy; Vascular Diseases; Cardiovascular Diseases; Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Renal Denervation (Experimental)
  Interventions: Device: Renal Denervation

INTERVENTIONS:
Device: Renal Denervation — Renal angiogram and renal denervation (Paradise ultrasound Renal Denervation System)

SUMMARY:
RADIANCE CAP is a non-randomized study designed to allow for continued access to ultrasound renal denervation therapy via the Paradise System, and to allow for the on-going collection of safety and effectiveness data in subjects with uncontrolled hypertension despite the prescription of antihypertensive medications.

ELIGIBILITY:
Inclusion Criteria:

* Average office BP ≥140/90 mmHg at screening visit despite taking stables doses of antihypertensive medications for at least 4 weeks prior to consent
* Documented daytime ABP ≥135/85 mmHg following 4 week run-in/standardization period on antihypertensive medication regimen

Exclusion Criteria:

* Renal artery anatomy ineligible for treatment
* Secondary hypertension not including sleep apnea
* Type I diabetes mellitus or uncontrolled Type II diabetes (defined as plasma HbA1c ≥9.0%)
* eGFR <40
* Brachial circumference ≥42 cm
* Any history of cerebrovascular event or severe cardiovascular event within 3 months prior to consent
* Documented repeat (>1) hospitalization for hypertensive crisis within 3 months prior to consent
* Documented confirmed episode(s) of unstable angina within 3 months prior to consent
* Chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea
* Primary pulmonary hypertension
* Night shift workers
* Pregnant, nursing or planning to become pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | From baseline to 60 months
Change in average daytime ambulatory systolic BP | From baseline to 2 months post procedure

SECONDARY OUTCOMES:
Change in average 24-hr/night-time ambulatory systolic BP | From baseline to 2 months post procedure
Change in average daytime/24-hr/night-time ambulatory systolic BP | From Baseline to Months 6 and 12 post procedure
Change in average office systolic/diastolic BP | From Baseline to Months 2, 6, 12, 24, 36, 48, and 60 post procedure
Change in average home systolic/diastolic BP | From Baseline to Months 2, 6, 12, 24, 36, 48, and 60 post procedure
Change in average 24-hr/night-time ambulatory diastolic BP | From baseline to Months 2, 6, and 12 post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Fisher, MD, Principal Investigator — Brigham and Women's Hospital/Harvard Medical School; Ajay Kirtane, MD, SM, Principal Investigator — Columbia University Medical Center/NYPH
Locations (40):
- United States (40):
  - Cardiovascular Institute of San Diego, Chula Vista, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sutter Health, Sacramento, California
  - Pacific Heart Institute, Santa Monica, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Emory, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - SIU Medicine, Springfield, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - UnityPoint Health-Des Moines, Des Moines, Iowa
  - Ochsner Medical Center, New Orleans, Louisiana
  - Lifebridge Health, Baltimore, Maryland
  - Tidal Health, Salisbury, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Luke's Hospital, Kansas City, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - NJ Heart & Vascular, Princeton, New Jersey
  - NYU Langone Hospital - Long Island, Mineola, New York
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cone Health, Greensboro, North Carolina
  - St. Francis Hospital, Tulsa, Oklahoma
  - Penn Medicine, Philadelphia, Pennsylvania
  - UPMC Heart and Vascular Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Texas Health Sciences Center at Houston, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - University of Texas Health Sciences Center, San Antonio, San Antonio, Texas
  - Baylor Scott & White Research Institute, Temple, Texas
  - Swedish Health Services, Seattle, Washington

REFERENCES:
- [Background] Azizi M, Sanghvi K, Saxena M, Gosse P, Reilly JP, Levy T, Rump LC, Persu A, Basile J, Bloch MJ, Daemen J, Lobo MD, Mahfoud F, Schmieder RE, Sharp ASP, Weber MA, Sapoval M, Fong P, Pathak A, Lantelme P, Hsi D, Bangalore S, Witkowski A, Weil J, Kably B, Barman NC, Reeve-Stoffer H, Coleman L, McClure CK, Kirtane AJ; RADIANCE-HTN investigators. Ultrasound renal denervation for hypertension resistant to a triple medication pill (RADIANCE-HTN TRIO): a randomised, multicentre, single-blind, sham-controlled trial. Lancet. 2021 Jun 26;397(10293):2476-2486. doi: 10.1016/S0140-6736(21)00788-1. Epub 2021 May 16. PMID 34010611
- See also: ReCor Medical company website — https://www.recormedical.com/
- See also: Study eligibility questionnaire; study summary and information — https://www.highbptrial.com